CLINICAL TRIAL: NCT03297190
Title: Evaluating the Impact of Text Messages and Interpersonal Community Support Groups on MICN Practices in Tanzania
Brief Title: Impact on Nutritional Practices: SMS and Interpersonal Communication
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Keller International (Other)
Collaborators: Tanzania Food and Nutrition Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 20171
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Nutritional Deficiency
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Four arms: (1) SMS only; (2) SMS + interpersonal; (3) interpersonal only; (4) none
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SMS (Active Comparator): Participants will receive SMS messages on nutrition and health related topics
  Interventions: Behavioral: SMS
- Interpersonal (Active Comparator): Participants will receive interpersonal counselling on nutrition and health related topics
  Interventions: Behavioral: Interpersonal Counselling
- SMS + Interpersonal (Active Comparator): Participants will receive SMS messages on nutrition and health related topics as well as interpersonal counselling on nutrition and health related topics
  Interventions: Behavioral: SMS; Behavioral: Interpersonal Counselling
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: SMS — Receipt of SMS messages on nutrition and health topics
  Arms: SMS; SMS + Interpersonal
Behavioral: Interpersonal Counselling — Interpersonal counselling on health and nutrition topics
  Arms: Interpersonal; SMS + Interpersonal

SUMMARY:
This cluster randomized controlled study aims to add to the evidence base on mHealth interventions by assessing the main effects of delivering nutrition messages on key maternal, infant, and young child nutrition (MIYCN) behaviors and outcomes through three innovative behavior change strategies. The strategies compared will be: (i) an interpersonal communication strategy using the Tanzanian government's Mkoba wa Siku 1000 maternal, infant and young child nutrition (MIYCN) curriculum (MwS) through clinic- and community-based channels, (ii) the mNutrition SMS text messaging module of the government's Wazazi Nipendeni program, and (iii) the combination of both of these strategies (interpersonal and SMS messaging). They will be compared with the current standard of care in Tanzania. The goal will be to determine which has the greatest impact on key MIYCN and hygiene practices and care-seeking behaviors. It will be paired with a costing analysis so that these effects can be understood in the context of their costs.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of children aged 0-12 mo. or pregnant at time of enrollment
* Consent to participate in the study

Exclusion Criteria:

* Unable to consent to participate in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2245 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Children's Dietary Diversity | 24 h
  % of children 6-29 mo. who consumed the minimum dietary diversity (received foods from ≥4 food groups on the previous day)
Women's dietary diversity | 24 h
  % who consumed food items from at least five out of ten defined food groups in the previous 24 hours (WDDS)
Children's Minimum Meal Frequency | 24 h
  % of children 6-29 mo. who consumed the minimum meal frequency the prior day (2/day for breastfed infants 6-8 mo.; 3/day for breastfed infants 9-29 mo.; 4/day for non-breastfed infants 6-29 mo.)

CONTACTS AND LOCATIONS:
Locations (1):
- HKI-Tanzania, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data to be shared after data analysis is completed.
Supporting Information: Study Protocol, ICF
Time Frame: Approximately 12 mo. after completion, indefinitely
Access Criteria: Fill out data use agreement.